CLINICAL TRIAL: NCT05696522
Title: Stereotactic Ablative Radiotherapy for the Treatment of Refractory Ventricular Tachycardia
Acronym: SABRE-VT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 262246
Record Dates: First submitted 2022-02-21; First posted 2023-01-25 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Radiotherapy; Complications; Ventricular Tachycardia; Structural Heart Abnormality; Heart Failure
Keywords: radiotherapy; ventricular tachycardia; heart failure
MeSH Terms: conditions — Tachycardia, Ventricular; Heart Failure

STUDY DESIGN:
Intervention Model Description: Prospective, interventional, pilots study with open label, non-randomised design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Treatment with stereotactic ablative radiotherapy
  Interventions: Radiation: Stereotactic ablative radiotherapy

INTERVENTIONS:
Radiation: Stereotactic ablative radiotherapy — Stereotactic ablative radiotherapy will be delivered to a volume of ventricular myocardium responsible for the clinical ventricular tachycardia.

SUMMARY:
Ventricular tachycardia (VT) is an abnormal rhythm arising from the bottom chambers (ventricles) of the heart. The hearts of most patients who develop VT have been previously damaged by a myocardial infarction (heart attack) or other heart muscle diseases (cardiomyopathies). The damage produces scar or fatty deposits that conduct electrical impulses slowly allowing VT to occur. Recurrent episodes of VT can compromise heart function and increase mortality.

VT is prevented by special drugs but these are not always effective and can have many side effects. Most patients with VT will also have a specialised device called an implantable defibrillator (ICD) implanted. The ICD treats VT by either stimulating the heart rapidly or delivering a shock to it. ICDs are very effective but the shocks are painful and have a big impact on quality of life. If VT occurs despite optimal drug treatment, patients undergo an invasive procedure called catheter ablation. Here, wires are passed into the heart from the blood vessels in the leg and the damaged heart muscle causing the VT is identified whilst the heart is in VT. An electrical current is passed down the wire making its tip heat up allowing discrete burns (ablation) to be placed inside the heart. The ablated heart muscle doesn't conduct electricity which stops the VT and prevents it recurring.

Some patients are so frail that ablation cannot be performed safely. A recent clinical trial has shown that VT can be treated in such patients using radiotherapy, which is usually used to treat tumours with high energy radiation. This approach is non-invasive, painless and requires no sedation or anaesthesia.

This study will test whether VT can be successfully treated using stereotactic ablative radiotherapy. This can deliver high dose radiotherapy very precisely, whilst minimising the risk of damage to healthy tissues.

DETAILED DESCRIPTION:
Principal objectives:

1. To determine the safety and efficacy of stereotactic ablative radiotherapy (SABR) for the treatment of VT refractory to conventional therapies.

Background:

VT is an abnormal heart rhythm arising from either of the bottom chambers of the heart (ventricles). Most patients with VT have scarring or fatty deposits in the heart muscle caused by a previous heart attack or a heart muscle problem called a cardiomyopathy. The abnormal heart muscle conducts electricity slowly allowing VT to occur. Most patients with VT have a device called an implantable defibrillator (ICD) fitted to treat VT. The ICD has wires going into the heart from a small generator that is inserted under the skin below the left collar bone. ICDs stop VT by stimulating the heart rapidly or by shocking the heart which is very painful and can stun the heart temporarily, weakening its pumping function. Patients who experience a lot of VT can have more admissions to hospital, worsening heart failure and a poorer quality of life, as well as a higher risk of dying. Consequently, all patients are treated with drugs to prevent VT but these are not always effective. If VT keeps recurring, many patients undergo an invasive procedure called catheter ablation where wires are passed into the heart from the leg and the part of the ventricles causing the VT identified. A high frequency electrical current is then passed down one of the wires making its tip heat up allowing discrete burns (ablation) to be placed on the culprit area, which stops the VT and prevents it from recurring. Performing catheter ablation in such patients is a high risk procedure and the overall complication rate is between 5 - 15% in experienced centres. Some patients have recurrent VT despite catheter ablation or the VT cannot be ablated because the patient is too frail, or the VT causes a significant fall in the blood pressure resulting in cardiac arrest (heart stops beating).

In the last 6 years, several case reports and series have been published showing that radiotherapy using different types of linear accelerator machines (including the Cyberknife) can successfully and safely ablate VT. Most recently, a prospective, randomised trial (ENCORE-VT) has reported a dramatic reduction in VT following radioablation.

This study will therefore assess our ability to perform stereotactic radioablation for VT at St Bartholomew's Hospital. We will determine procedural success and safety. Patients will be assessed 3, 6 and 12 months after the treatment and their burden of VT determined by checking the ICD.

ELIGIBILITY:
Inclusion Criteria:

1. They are at least 18-85 years old.
2. They have recurrent VT (at least three episodes in the preceding six months) requiring therapy from an ICD, that is refractory to conventional treatments - both maximally tolerated doses of anti- arrhythmic drugs and/or conventional catheter ablation.
3. They are too frail or do not wish to undergo conventional catheter ablation.
4. They have not had previous radiotherapy to the anticipated treatment field.

Exclusion Criteria:

1. They have polymorphic VT or ventricular fibrillation (VF).
2. They have inotrope-dependent heart failure or a left ventricular assist device (LVAD) in situ.
3. They are unlikely to live more than 12 months irrespective of the VT.
4. There is a potentially reversible cause for the VT e.g. critical coronary artery disease or a metabolic problem such as an overactive thyroid gland.
5. They are unable to provide informed consent.
6. They have had previous radiotherapy to the anticipated treatment field.
7. The patient weighs in excess of 170kg (maximum weight capacity of the tables in the imaging department).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2026-05-02 (Estimated); Study Completion 2026-05-02 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life and cardiac complications as assessed by clinical history, SF-36 questionnaire, electrocardiogram and echocardiography. | 3 months
  The number of serious adverse events at three months after treatment. This will be determined as follows:
  1. Clinical history from and examination of the patients assessing for new chest pains, breathlessness or coughing.
  2. SF-36 quality of life questionnaire.
  3. Echocardiography to assess for pericardial effusion that could indicate radiation-induced pericarditis.
  4. Electrocardiogram to assess for pericarditis or myocarditis caused by radiation.
Efficacy endpoint - Cumulative VT burden 6 months before and 6 months after radiotherapy. | 6 months
  There will be a six week blanking period after radiotherapy to allow for ablation effect. The burden of VT will be assessed by interrogating the patient's ICD and assessing the number of episodes of non-sustained and sustained VT as well as the number of ICD therapies delivered.

SECONDARY OUTCOMES:
VT burden | 6 months
  Cumulative VT burden in the second 6 months following radiotherapy. This will be assessed by ICD interrogation as described above.
Survival | 12 months
  Overall survival at 3, 6 and 12 months following radiotherapy.
Cardiac function changes from radiotherapy | 12 months
  Absolute change in numerical left ventricular ejection fraction assessed with echocardiography, at 3, 6 and 12 months.
Radiotherapy impact on ICD function | 12 months
  Deterioration in implantable cardioverter-defibrillator function attributable to radiotherapy at 3, 6 and 12 months. This will be determined by interrogating the ICD and measuring the change in ICD defibrillator lead impedance.
Quality of life assessment using SF-36 questionnaire | 12 months
  The SF-36 questionnaire will be used at 3, 6 and 12 months to assess this.
Heart failure status using New York Heart Association (NYHA) breathlessness class. | 12 months
  Patients will be assessed at 3, 6 and 12 months by taking a history for breathlessness, scaled I to IV according to their NYHA class.
Cardiac conduction system status measured by ECG QRS duration. | 12 months
  An electrocardiogram will be performed at 3, 6 and 12 months to look for any changes in the QRS complex duration.

CONTACTS AND LOCATIONS:
Locations (1):
- St Bartholomew's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No